CLINICAL TRIAL: NCT01290627
Title: In Vivo Determination of 3D Patellofemoral Mechanics
Acronym: Patella
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: 10035/IIS-000126; R011373372 (Other Grant/Funding Number: DePuy Orthopaedics)
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Arthroplasty Replacement Knee; Knee Prosthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Knee Prosthesis LCS PS RP TKA: Subjects implanted with DePuy Low Contact Stress (LCS) Poster Stabilizing (PS) Rotating Platform (RP) Total Knee Arthroplasty (TKA)
  Interventions: Device: Subjects implanted with DePuy LCS PS RP TKA
- Knee Prosthesis Sigma PS RP TKA: Subjects implanted with a DePuy Sigma Posterior Stabilizing (PS) Rotating Platform (RP) Total Knee Arthroplasty (TKA)
  Interventions: Device: Subjects implanted with DePuy Sigma PS RP TKA
- Control: Subjects with normal knees

INTERVENTIONS:
Device: Subjects implanted with DePuy LCS PS RP TKA — Subjects implanted with DePuy Low Contact Stress (LCS) Poster Stabilizing (PS) Rotating Platform (RP) Total Knee Arthroplasty (TKA)
  Groups: Knee Prosthesis LCS PS RP TKA
Device: Subjects implanted with DePuy Sigma PS RP TKA — Subjects implanted with a DePuy Sigma Posterior Stabilizing (PS) Rotating Platform (RP) Total Knee Arthroplasty (TKA)
  Groups: Knee Prosthesis Sigma PS RP TKA

SUMMARY:
This study will analyze the tibio-femoral and patellofemoral (motion) and mechanics (forces) of participants having a normal knee or a total knee arthroplasty (TKA) using one or two different (TKA) devices Low Contract Stress (LCS) Posterior Stabilizing (PS) Rotating Platform (RP) Total Knee Arthroplasty (TKA). All knees will be analyzed using an image matching technique that will convert a two-dimensional (2D) fluoroscopic image into a three-dimensional (3D) image. In conjunction with the fluoroscopic analysis, electromyography (EMG) data, and ground reaction force (GRF) data will all be allow for a complete analysis of the knee joints. These results will help the orthopaedic community better understand knee motion so they can improve testing on existing implants and develop future implants that will further enhance patients' lives.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least six months post-operative.
2. Potential subjects will have a body weight of less than 250 lbs.
3. Candidates must have an AKS score >70 post-operatively.
4. Patients must have passive flexion of at least 100.
5. Implanted group must have either an LCS PS RP TKA, having an anatomical patella, or Sigma PS RP TKA; or normal knee group must have normal knee.
6. Must be willing to sign both Informed Consent and HIPAA forms.

Exclusion Criteria:

1. Pregnant females.
2. Subjects not meeting study requirements.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects recruited from patients chosen from practice of Dr.'s Dennis and Haas at Colorado Joint Replacement for implanted knee, having either one of the two kinds of implants specified.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Komistek, Ph D, Principal Investigator — The University of Tennessee; Douglas Dennis, MD, Principal Investigator — Colorado Joint Replacement, Porter Adventist Hosp
Locations (4):
- United States (4):
  - Colorado Joint Replacement, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Perkins Hall, Knoxville, Tennessee
  - Science and Engineering Research Facility, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Colorado Joint Replacement practice of Drs. Doug Dennis and Brian Haas in Denver, CO after the study was approved by respective IRBs beginning 5/27/11.
Period: Overall Study
Arm/Group | Knee Prosthesis LCS PS RP TKA | Knee Prosthesis Sigma PS RP TKA | Control
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Knee Prosthesis LCS PS RP TKA | Knee Prosthesis Sigma PS RP TKA | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10 | 20
  >=65 years | 5 | 5 | 0 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (7.8) | 64.3 (8.7) | 34.2 (8.9) | 53.67 (16.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 8 | 13
  Male | 6 | 9 | 2 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Patella Flexion With Respect to Femur
Description: Full extension to maximum flexion. Degrees of flexion analyzed for participants with and without implants.
Time Frame: Average post-operative time for LCS-PS group was 56 months. Average post-operative time for PS RP group was 55.7 months.
Population: Unit analyzed is an orthopaedic implant and subjects with normal knees do not have orthopaedic implants.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Implants/Knees
Arm/Group | Knee Prosthesis LCS PS RP TKA | Knee Prosthesis Sigma PS RP TKA | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (Implants/Knees) | 10 | 10 | 10
degrees | 80.0 (13.6) | 83.4 (12.9) | 93.7 (12.9)

2. Primary Outcome: Patella Rotation With Respect to Femur
Description: Patellar rotation from full extension to maximum flexion for subjects with and without implants. A positive measurement of patellar rotation refers to positive flexion of the patella about the medial-lateral axis, where the patella component rotates so that the top of the patella rotates toward the femur and the bottom rotates away. Conversely, a negative measurement refers to negative flexion of the patella about this axis, where the patellar component rotates so that the top of the patella moves away from the femur and the bottom moves towards.
Time Frame: Average post-operative time for LCS-PS group was 56 months. Average post-operative time for PS RP group was 55.7 months.
Population: Unit analyzed is an orthopaedic implant and subjects with normal knees do not have orthopaedic implants.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Implants/Knees
Arm/Group | Knee Prosthesis LCS PS RP TKA | Knee Prosthesis Sigma PS RP TKA | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (Implants/Knees) | 10 | 10 | 10
degrees | .5 (5.0) | -.06 (3.1) | -1.6 (6.1)

3. Primary Outcome: Patella Tilt With Respect to Femur
Description: full extension to maximum flexion for participants with and without implants.
Time Frame: Average post-operative time for LCS-PS group was 56 months. Average post-operative time for PS RP group was 55.7 months.
Population: Unit analyzed is an orthopaedic implant and subjects with normal knees do not have orthopaedic implants.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Implants/Knees
Arm/Group | Knee Prosthesis LCS PS RP TKA | Knee Prosthesis Sigma PS RP TKA | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (Implants/Knees) | 10 | 10 | 10
degrees | 4.2 (5.1) | 2.6 (6.4) | 5.3 (5.9)

4. Primary Outcome: Normalized Medial Patella Contact Point Translation
Description: full extension to maximum flexion for participants with and without implants. Position of the patellar contact point was determined by locating the closest point to the femur on the patella throughout flexion. There are 2 patello-femoral contact points: a point on the medial aspect of the patella and a point on the lateral aspect of the patella. Throughout flexion, the medial contact point generally moves closer to the top of the patella (hence the positive value for the results). The translation of this contact point is normalized to report a ratio between -1 and 1. In other words, the distance the point has traveled compared to the total height of the patella. For example, if the patella is 8 cm in height and the point travels approximately 2 cm upwards during flexion, the value would be reported as +2/8 = +0.25. Definition of normalized: "multiply (a series, function, or item of data) by a factor that makes the norm or some associated quantity such as an integral equal
Time Frame: Average post-operative time for LCS-PS group was 56 months. Average post-operative time for PS RP group was 55.7 months.
Population: Unit analyzed is an orthopaedic implant and subjects with normal knees do not have orthopaedic implants.
Measure: Mean (Standard Deviation); unit: ratio of patella height
Units Other Than Participants: Implants/Knees
Arm/Group | Knee Prosthesis LCS PS RP TKA | Knee Prosthesis Sigma PS RP TKA | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (Implants/Knees) | 10 | 10 | 10
ratio of patella height | .34 (.18) | .12 (.17) | .40 (.41)

5. Primary Outcome: Normalized Lateral Patella Contact Point Translation
Description: full extension to maximum flexion for participants with and without implants. Position of patellar contact point was determined by locating closest point to femur on patella throughout flexion. There are 2 patello-femoral contact points: 1 point on the medial aspect of the patella and 1 point on the lateral aspect of the patella. Throughout flexion, lateral contact point generally moves closer to the top of the patella (hence, the positive value for the results). The translation of this contact point is normalized to report a ratio between -1 and 1. The distance the point has traveled compared to the total height of the patella. For example, if the patella is 8 cm in height and the point travels approximately 2 cm upwards during flexion, the value would be reported as +2/8 = +0.25. Definition of normalized: "multiply (a series, function, or item of data) by a factor that makes the norm or some associated quantity such as an integral equal to a desired value (usually 1)."
Time Frame: Average post-operative time for LCS-PS group was 56 months. Average post-operative time for PS RP group was 55.7 months.
Population: Unit analyzed is an orthopaedic implant and subjects with normal knees do not have orthopaedic implants.
Measure: Mean (Standard Deviation); unit: ratio of patella height
Units Other Than Participants: Implants/Knees
Arm/Group | Knee Prosthesis LCS PS RP TKA | Knee Prosthesis Sigma PS RP TKA | Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (Implants/Knees) | 10 | 10 | 10
ratio of patella height | 0.09 (.22) | .20 (.17) | .45 (.52)

ADVERSE EVENTS:
Description: There were no adverse effects or events encountered for any subjects in this study.
Arm/Group | Knee Prosthesis LCS PS RP TKA | Knee Prosthesis Sigma PS RP TKA | Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
No adverse effects, events or unexpected risks occurred The sample size per group was small Age of the TKA groups were matched, the age of the normal subjects were not Cartilage thickness for normals had to be assumed as MRIs could not be obtained

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No